CLINICAL TRIAL: NCT04623307
Title: Clinical Applications for Non-contact DCS-Speckle Multi-parameter Imaging for Brain Injuries and Brain Edema
Brief Title: Non-contact DCS-Speckle Multi-parameter Imaging for Neurological Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ting Li (Unknown)
Collaborators: Beijing Geriatric Hospital (Other); Tianjin Huanhu Hospital (Other)
Responsible Party: Sponsor-Investigator, Ting Li, Full professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: Brain disease for DCS-Speckle
Record Dates: First submitted 2020-11-09; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Brain Injuries; Brain Edema; Optical Imaging
Keywords: DCS-Speckle; Brain injuries; Brain edema
MeSH Terms: conditions — Brain Injuries; Brain Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Brain damage patients: Brain damage patients were monitored the human brain activity by the non-contact DCS-Speckle multi-parameter imager.
  Interventions: Diagnostic Test: Non-contact DCS-Speckle multi-parameter imaging
- Brain edema patients: Brain edema patients were monitored the human brain activity by the non-contact DCS-Speckle multi-parameter imager.
  Interventions: Diagnostic Test: Non-contact DCS-Speckle multi-parameter imaging
- Healthy subjects: Healthy subjects were monitored the human brain activity by the non-contact DCS-Speckle multi-parameter imager.
  Interventions: Diagnostic Test: Non-contact DCS-Speckle multi-parameter imaging

INTERVENTIONS:
Diagnostic Test: Non-contact DCS-Speckle multi-parameter imaging — The protocol consists of 2-min resting, 6-min stationary state and 2-min resting, with monitoring data continuously by the DCS-Speckle.

SUMMARY:
This study aims to evaluate brain injuries and brain edema with non-contact DCS-Speckle multi-parameter imager.

DETAILED DESCRIPTION:
Brain injuries includes acute and chronic injuries located in cerebral hemispheres, cerebellum, and brain stem, while brain edema is increased intracellular or extracellular fluid in brain tissue. Early diagnosis is helpful to improve the cure rate and reduce sequelae. This study aims to evaluate brain injuries and brain edema with non-contact DCS-Speckle multi-parameter imager, so as to provide reference diagnostic criteria by image artificial intelligence analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had brain damage.
* Patients who have had brain edema.
* Healthy people who are interested in non-contact DCS-Speckle multi-parameter imaging

Exclusion Criteria:

* Patients who are in pregnancy or have plan to conception.
* Patients who have vertebra surgery or have plan to surgery.
* Patients who are inappropriate to join this trial judged by the radiologists or specialists.
* AIDS, Active Hepatitis, Tuberculosis, Syphilis
* Patients who regularly take anticoagulants, antiplatelet drugs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult individuals and infants of any gender. Brain damage patients were hired in Beijing Geriatric Hospital, and brain edema patients hired in Tianjin Huanhu Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging data | 1 day during the whole experiment
  Imaging data collected during the non-contact DCS-Speckle imaging instrument

SECONDARY OUTCOMES:
Diagnostic report fMRI data | 1 day during the whole experiment
  Patients' medical record and diagnostic report

CONTACTS AND LOCATIONS:
Locations (1):
- NIRS assessment for brain death, Tianjin, Tianjin Municipality, China